CLINICAL TRIAL: NCT04335266
Title: A Randomized, Open, Single-center, Two-cycle, Double-sequence Crossover Study to Investigate the Effects of a High-fat Diet on the Pharmacokinetics of Healthy Chinese Male Adult Subjects After Oral Administration of SHR2554 Tablets
Brief Title: A Food Effect Study of SHR2554 on Healthy Chinese Male Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SHR2554-I-103
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): Drug: SHR2554 fasted in P1, high-fat diet in P2 SHR2554 administration in fasted condition in period 1, SHR2554 administration after high-fat diet in period 2
  Interventions: Drug: SHR2554
- Treatment group B (Experimental): Drug: SHR2554 high-fat diet in P1, fasted in P2 SHR2554 administration after high-fat diet in period 1, SHR2554 administration in fasted condition in period 2
  Interventions: Drug: SHR2554

INTERVENTIONS:
Drug: SHR2554 — SHR2554

SUMMARY:
The primary objective of the study is to evaluate the effect of high-fat diet on pharmacokinetics of healthy Chinese male adult subjects after oral administration of SHR2554 tablets.

The secondary objective of the study is to evaluate the safety of single dose of SHR2554 orally in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 40~60 at the date of signing the informed consent;
2. Male body weight ≥ 50kg , body mass index (BMI) within the range of 19 ~ 28kg /m2 (including 19 and 28) (BMI= weight (kg)/height 2 (m2));
3. During screening period physical examination, vital signs, blood routine, urine routine, blood biochemistry, coagulation, abdominal ultrasound, chest X-ray and other examination results must be within the normal range consistent with age and gender, or in accordance with the protocol, or judged to be "no clinical significance (NCS)" if beyond the normal range;
4. Agree to abstain from sex or use effective non-drug contraceptives from screening to at least 3 months after the last study drug administration (female subjects are also required to abstain or use effective non-drug contraceptives two weeks prior to study entry);
5. The subject can communicate well with the researcher, understand and comply with the requirements of the study, understand and sign the informed consent.

Exclusion Criteria:

1. Allergic constitution or known allergy to the research drug/similar drugs;
2. Frequent use of sedatives, sleeping pills or other addictive drugs; History of drug abuse within 6 months prior to first administration or drug abuse screening positive; Alcoholic or often drinkers within 6 months prior to screening, the average drinking amount is more than 14 units a week (1 unit= 285 ml beer or 25 ml alcohol content of 40% spirits or 100 ml wine), a heavy smoker or quitting time less than 3 months, alcohol breath test positive and nicotine test positive, and can't quit smoking and alcohol during the study;
3. A history of cardiovascular diseases such as myocarditis, coronary heart disease, pathological arrhythmia and stroke;
4. Pulmonary diseases, including invasive lung disease, pneumonia, and dyspnoea;
5. Chronic kidney disease, renal insufficiency, renal anaemia;
6. A history of dysphagia or any gastrointestinal disease affecting drug absorption;
7. Any uncontrolled peptic ulcer, colitis, pancreatitis, etc;
8. Any operation within the previous 3 months that may affect the absorption, distribution, metabolism and excretion of drugs;
9. Previous medical history of cardiovascular, liver, kidney, lung, digestive tract, nervous system diseases, etc., which may significantly affect the absorption, distribution, metabolism and excretion of drugs, or may pose a hazard to the subjects participating in the study. The following medical history or conditions should be considered: inflammatory gastroenteritis, gastroesophageal reflux, gastrointestinal or rectal bleeding; History of pancreatic injury or pancreatitis; Greater surgical history such as gastrectomy, gastroenterostomy, or enterectomy; History of acute and chronic renal insufficiency, history of renal transplantation;
10. Taking any hepatotoxic drugs (such as dapsone, erythromycin, fluconazole, ketoconazole and rifampicin) in the months prior to screening;
11. hose who have participated in other clinical trials and taken the research drugs within 3 months before the first drug administration;
12. Any drug that altered the activity of liver enzymes was given 28 days prior to administration or during the study;
13. Use any prescription drug or herbal tonic within one week before the first dose;
14. Use any over-the-counter (OTC) or food supplement (including vitamins, calcium tablets, etc.) within one weeks before the first dose;
15. Clinical laboratory examination is abnormal and to be CS;
16. Hepatitis B surface antigen positive, hepatitis C2 antibody positive, syphilis antibody positive, HIV antibody positive;
17. Subjects refused to stop using any beverage or food containing methyl xanthine, such as coffee, tea, cola, chocolate, etc. from 48 hours before the first administration until the end of the study;
18. Blood donation within 3 months before the screening or blood loss great than 400 mL;
19. Difficulty in venous blood collection or inability to tolerate venepuncture;
20. Other factors (including but not limited to inability to understand the requirements of the study, poor compliance, physical weakness, etc.) that are not suitable for participating in the study, as judged by the researcher.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of SHR2554 | Day 1 and Day 8 of the single dose
  Peak Plasma Concentration (Cmax) of SHR2554
Pharmacokinetics parameter: AUC of SHR2554 | Day 1 and Day 8 of the single dose
  Area under the plasma concentration versus time curve (AUC) of SHR2554

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Henan, China

IPD SHARING:
Plan to Share IPD: No